CLINICAL TRIAL: NCT03579186
Title: Optokinetic Stimulation for the Treatment of Gait Abnormalities
Brief Title: OKS for Gait Instability
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment and other trial activities have temporarily paused due to COVID-19 and are expected to resume in the future; This is not a suspension of IRB approval
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Chun Lim, Assistant Professor, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2015P000091
Record Dates: First submitted 2018-03-21; First posted 2018-07-06 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2021-08

CONDITIONS: Gait, Unsteady; Vestibular Disorder
MeSH Terms: conditions — Gait Disorders, Neurologic; Vestibular Diseases

STUDY DESIGN:
Intervention Model Description: Patients undergoing a clinical gait assessment will be recruited for this study. Those that consent to participate will complete their clinical gait assessment as part of their normal evaluation. Subjects will then complete a gait assessment while wearing experiencing optokinetic stimulation. The investigators will compare baseline gait and postural control before and during OKS stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait (Experimental): Patients undergoing a routine clinical gait assessment at the Brain Fit Club at BIDMC will have their posture and gait measured before and during optokinetic stimulation (OKS).
  Interventions: Device: OKS

INTERVENTIONS:
Device: OKS — Optokinetic stimulation

SUMMARY:
Specific aim: To determine whether optokinetic stimulation can improve gait abnormalities.

Hypothesis: Optokinetic stimulation stimulates the vestibular system and can improve vestibular induced gait disorders.

DETAILED DESCRIPTION:
This is a pilot study designed to determine whether or not the optokinetic stimulation improves gait in patients with gait abnormalities, specifically vestibular induced gait disorders. The study population will consist of patients already receiving a gait assessment through the Brain Fit Club (BFC) at Beth Israel Deaconess Medical Center. This gait assessment involves walking and posture evaluations. Patients will complete a gait assessment as part of their normal BFC evaluation. Those who consent to participate in the study will then complete a gait assessment while receiving optokinetic stimulation. The investigators will compare baseline gait and postural control before and during OKS stimulation.

ELIGIBILITY:
Inclusion criteria:

* Receiving a gait assessment through the BFC
* Ages 21-75

Exclusion criteria:

* Left hemiparesis
* Requires a cane or walker
* Documented evidence of falls or instability to the left
* Reduced vision
* Moderate or severe dementia

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Gait - (measured using a wireless 3D accelerometer) | After 5 minutes of OKS
  Change in walking balance (lateral step deviation) as measured using a wireless 3D accelerometer
Posture - (measured using a stationary force platform) | After 5 minutes of OKS
  Change in standing balance (left-right deviation) as measured using a stationary force platform.

SECONDARY OUTCOMES:
Speed | After 5 minutes of OKS
  Change in gait speed

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No